CLINICAL TRIAL: NCT01175824
Title: Comparison of Twice-Daily Insulin Lispro Low Mixture Versus Once-Daily Basal Insulin Glargine and Once-Daily Prandial Insulin Lispro as Insulin Intensification Strategies in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Basal Insulin Glargine and Metformin and/or Pioglitazone
Brief Title: Comparison of the Efficacy and Safety of Two Insulin Intensification Strategies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13493; F3Z-CR-IOQE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metabolic Diseases; Diabetes Mellitus, Type 2; Glargine; Diabetes Mellitus; Insulin LISPRO; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Diseases; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin lispro low mixture (LM) (Experimental): Two daily injections (breakfast and dinner) of insulin lispro mix 75/25
  Interventions: Drug: Insulin Lispro Low Mixture (LM)
- Insulin glargine+insulin lispro (Active Comparator): Once-daily (bedtime) basal insulin glargine and once-daily (before the main meal with the highest average 2-hour postprandial blood glucose concentration) prandial insulin lispro
  Interventions: Drug: Insulin Glargine; Drug: Prandial Insulin Lispro

INTERVENTIONS:
Drug: Insulin Lispro Low Mixture (LM) — Participant-dependent dose, administered subcutaneously for 24 weeks
  Other Names: Humalog Mix75/25 (75% insulin lispro protamine suspension and 25% insulin lispro injection)
  Arms: Insulin lispro low mixture (LM)
Drug: Insulin Glargine — Participant-dependent dose, administered subcutaneously for 24 weeks
  Arms: Insulin glargine+insulin lispro
Drug: Prandial Insulin Lispro — Participant-dependent dose, administered subcutaneously for 24 weeks
  Other Names: Humalog; LY275585
  Arms: Insulin glargine+insulin lispro

SUMMARY:
The study is a comparison of twice-daily insulin lispro low mixture versus once-daily basal insulin glargine and once-daily prandial insulin lispro, in participants with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Present with type 2 diabetes mellitus
* Have been taking metformin and/or pioglitazone
* Have received treatment with basal insulin glargine, injected once a day, for greater than or equal to 90 days
* Have glycosylated hemoglobin A1c (HbA1c) concentration between greater than or equal to 7.5% and less than or equal to 10.5
* Have a fasting plasma glucose concentration of less than or equal to 6.7 millimoles per liter [mmol/L, less than or equal to 121 milligrams per deciliter (mg/dL)], or greater than 6.7 mmol/L (greater than 121 mg/dL) if the investigator considers that further titration of basal insulin glargine is not possible for safety reasons
* Not pregnant or breastfeeding

Exclusion Criteria:

* Have Type 1 Diabetes
* Their stable dose of pioglitazone is greater than the maximum dose approved for use in combination with insulin in their country
* Have a body mass index (BMI) greater than 45 kilograms per square meter (kg/m2).
* Have a history of scheduled mealtime (prandial) insulin use within 12 weeks of the screening visit and the total duration of the prandial insulin treatment was greater than 2 weeks
* Have had more than one episode of severe hypoglycaemia within 24 weeks prior to entry into the study
* Have cardiac disease with a functional status that is Class III or IV
* Have a history of renal or liver disease
* Have had a blood transfusion or have a blood disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramos Mejía
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- China (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
- Egypt (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairo
- India (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Visakhapatnam
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyunggi-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Boi de Llobregat
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul

REFERENCES:
- [Derived] Rojas A, Sposetti G, Gross JL, Barbieri DE, Duan R, Linetzky B, De Lana JM, Stempa O, Rodriguez A. Insulin lispro low mixture twice daily vs basal insulin glargine once daily and prandial insulin lispro once daily as insulin intensification strategies in patients with type 2 diabetes: Latin American subpopulation analysis of a randomized trial. Diabetol Metab Syndr. 2016 Sep 17;8:69. doi: 10.1186/s13098-016-0163-3. eCollection 2016. PMID 27660663
- [Derived] Gross JL, Rojas A, Shah S, Tinahones FJ, Cleall S, Rodriguez A. Efficacy and safety of a premixed versus a basal-plus insulin regimen as intensification for type 2 diabetes by timing of the main meal. Curr Med Res Opin. 2016 Jun;32(6):1109-16. doi: 10.1185/03007995.2016.1161609. Epub 2016 Apr 7. PMID 26934128
- [Derived] Tinahones FJ, Gross JL, Onaca A, Cleall S, Rodriguez A. Insulin lispro low mixture twice daily versus basal insulin glargine once daily and prandial insulin lispro once daily in patients with type 2 diabetes requiring insulin intensification: a randomized phase IV trial. Diabetes Obes Metab. 2014 Oct;16(10):963-70. doi: 10.1111/dom.12303. Epub 2014 May 6. PMID 24725616

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Lispro Low Mixture: Two daily injections (breakfast and dinner) of insulin lispro mix 75/25. Participant-dependent doses, administered subcutaneously for 24 weeks.
- Insulin Glargine+Insulin Lispro: Once-daily injection (bedtime) basal insulin glargine and once-daily injection (before the meal with the highest average 2-hour postprandial blood glucose concentration) prandial insulin lispro. Participant-dependent doses, administered subcutaneously for 24 weeks.
Period: Overall Study
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Started | 236 | 242
Received at Least 1 Dose of Study Drug | 236 | 240
Completed | 220 | 220
Not Completed | 16 | 22
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 4
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Sponsor Decision | 1 | 0
Not completed — Entry Criteria Not Met | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: randomized participants who received at least 1 dose of study drug. Participants were analyzed per the assigned treatment arm regardless of the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro | Total
Number analyzed (Participants) | 236 | 240 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.93) | 57.7 (9.12) | 57.5 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 142 | 262
  Male | 116 | 98 | 214
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 15 | 17 | 32
  Asian | 80 | 80 | 160
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 133 | 136 | 269
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 40 | 39 | 79
  Brazil | 20 | 23 | 43
  China | 15 | 13 | 28
  Egypt | 5 | 7 | 12
  India | 40 | 41 | 81
  Korea, Republic of | 25 | 26 | 51
  Mexico | 20 | 20 | 40
  Romania | 38 | 38 | 76
  Russian Federation | 2 | 3 | 5
  Spain | 23 | 23 | 46
  Turkey | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to 24 Weeks Endpoint (Per Protocol Population)
Description: The change from baseline to 24 weeks in the percentage of glycosylated hemoglobin A1c (HbA1c) in plasma. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included baseline HbA1c concentration as a covariate, treatment, country, week of visit, and treatment-by-week interaction as fixed effects, and participant and error as random effects.
Time Frame: Baseline, 24 weeks
Population: Per protocol population: randomized participants with the exception of participants who did not complete Week 24 visit, received study drug different from their randomized study treatment, violated any of the inclusion, exclusion, or discontinuation criteria, or were significantly noncompliant.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 220 | 216
percentage of HbA1c | -1.30 [-1.44 to -1.16] | -1.09 [-1.24 to -0.95]
Statistical Analysis 1: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Non-Inferiority or Equivalence — Non-inferiority will be concluded if the upper limit of the 95% confidence interval (CI) of the difference in the LS mean between the two treatment arms (twice-daily insulin lispro Low Mixture minus the comparator arm) at 24 weeks is <0.4%; LS mean difference = -0.21, 95% CI 2-sided [-0.38 to -0.04]

2. Secondary Outcome: Change in the HbA1c Concentration From Baseline to 12 Weeks Endpoint
Description: The change from baseline to 12 weeks in the percentage of glycosylated hemoglobin A1c (HbA1c) in plasma. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included baseline HbA1c concentration as a covariate, treatment, country, week of visit, and treatment-by-week interaction as fixed effects, and participant and error as random effects.
Time Frame: Baseline, 12 weeks
Population: Intention-to-treat population (ITT): randomized participants who received at least 1 dose of study drug and had HbA1c data at the 12 weeks. Participants were analyzed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 222 | 226
percentage of HbA1c | -1.12 [-1.26 to -0.98] | -1.01 [-1.15 to -0.87]
Statistical Analysis 1: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.1858, Mixed Models Analysis

3. Secondary Outcome: Number of Participants Who Achieve a Target HbA1c Concentration of Less Than 7% or Less Than or Equal to 6.5% at 24 Weeks
Time Frame: 24 weeks
Population: Intention-to-treat population (ITT): randomized participants who received at least 1 dose of study drug and had HbA1c data at 24 weeks. Participants were analyzed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 220 | 220
participants
  HbA1c <7% | 76 | 66
  HbA1c <=6.5% | 36 | 31
Statistical Analysis 1: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.3588, Fisher Exact — HbA1c concentration <7%
Statistical Analysis 2: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.5958, Fisher Exact — HbA1c <=6.5%

4. Secondary Outcome: Change in the Fasting Plasma Glucose Concentration From Baseline to 12 Weeks and 24 Weeks
Description: The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included baseline fasting plasma glucose value as a covariate, treatment, country, baseline HbA1c stratification level, week of visit, and treatment-by-week interaction as fixed effects, and participant and error as random effects.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Intention-to-treat population (ITT): randomized participants who received at least 1 dose of study drug and had fasting plasma glucose concentration data at the specified time points. Participants were analyzed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 222 | 222
millimoles per liter (mmol/L)
  Change at 12 Weeks (n= 222, 222) | 1.04 [0.67 to 1.41] | 0.64 [0.27 to 1.00]
  Change at 24 Weeks (n=219, 217) | 0.89 [0.52 to 1.27] | 0.75 [0.38 to 1.12]
Statistical Analysis 1: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.0827, Mixed Models Analysis — p-value is for the Week 12 comparison
Statistical Analysis 2: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.5353, Mixed Models Analysis — p-value is for the Week 24 comparison

5. Secondary Outcome: 7-point Self-Monitored Blood Glucose (SMBG) Profiles at 12 Weeks and 24 Weeks
Description: 7-point Self-monitored Blood Glucose (SMBG) Profiles are measures of blood glucose taken 7 times a day at the morning pre-meal, morning 2-hours post-meal, midday pre-meal, midday 2-hours post-meal, evening pre-meal, evening 2-hours post-meal, and 0300 hour [3 am]. Each participant took measures on 3 non-consecutive days and the average was calculated for each of the 7 time points. The mean of the 7-point averages was calculated for all the participants at baseline, Weeks 12 and 24. The least squares (LS) mean was estimated from mixed-effects model with repeated measures that included the baseline value of the variable as a covariate, treatment, country, baseline glycosylated hemoglobin A1c (HbA1c)stratification level, week of visit, and treatment-by-week interaction as fixed effects, and participant and error as random effects.
Time Frame: 12 weeks, 24 weeks
Population: Intention-to-treat population (ITT): randomized participants who received at least 1 dose of study drug and had SMBG data at the specified time points. Participants were analyzed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 229 | 235
millimoles per liter (mmol/L)
  pre-morning meal (Week 12) (n=223, 222) | 6.87 [6.67 to 7.07] | 6.20 [6.01 to 6.40]
  2 hour post-morning meal (Week 12) (n=220, 221) | 8.82 [8.50 to 9.13] | 9.01 [8.70 to 9.33]
  pre-midday meal (Week 12) (n=220, 221) | 6.96 [6.68 to 7.24] | 7.44 [7.17 to 7.72]
  2 hours post-midday meal (Week 12) (n=220, 221) | 9.46 [9.14 to 9.78] | 9.14 [8.83 to 9.45]
  pre-evening meal (Week 12) (n=221, 221) | 7.98 [7.69 to 8.28] | 8.25 [7.96 to 8.54]
  2 hours post-evening meal (Week 12) (n=217, 220) | 9.15 [8.79 to 9.52] | 9.10 [8.74 to 9.46]
  3 am - during the night (Week 12)(n=197, 201) | 8.21 [7.87 to 8.55] | 8.52 [8.19 to 8.86]
  pre-morning meal (Week 24) (n=217, 216) | 6.60 [6.41 to 6.79] | 6.26 [6.07 to 6.45]
  2 hours post-morning meal (Week 24) (n=216, 215) | 8.52 [8.22 to 8.83] | 8.86 [8.56 to 9.16]
  pre-midday meal (Week 24) (n=215, 216) | 6.82 [6.54 to 7.09] | 7.44 [7.17 to 7.71]
  2 hours post-midday meal (Week 24) (n=216, 216) | 9.08 [8.76 to 9.40] | 8.99 [8.68 to 9.30]
  pre-evening meal (Week 24) (n=216, 216) | 7.70 [7.41 to 7.99] | 7.95 [7.66 to 8.24]
  2 hours post-evening meal (Week 24) (n=212, 216) | 9.11 [8.76 to 9.47] | 8.95 [8.60 to 9.30]
  3 am - during the night (Week 24)(n=198, 195) | 8.05 [7.72 to 8.38] | 8.26 [7.93 to 8.59]

6. Secondary Outcome: Glycemic Variability From the 7-point Self-Monitored Blood Glucose (SMBG) Profiles at 12 Weeks and 24 Weeks
Description: The 7-point SMBG profile was calculated as the average blood glucose concentration across the 7 pre-specified time points in a day that was then averaged over 3 non-consecutive days in the 2 weeks prior to the 12 week visit and 24 week visit. Glycemic variability was calculated as the standard deviation of the 7-point SMBG profiles. Standard deviation was first calculated for each day and then averaged over 3 non-consecutive days for each visit. The least squares (LS) mean was estimated from mixed-effects model with repeated measures that included the baseline value of the variable as a covariate, treatment, country, baseline glycosylated hemoglobin A1c (HbA1c)stratification level, week of visit, and treatment-by-week interaction as fixed effects, and participant and error as random effects.
Time Frame: 12 weeks, 24 weeks
Population: Intention-to-treat population (ITT): randomized participants who received at least 1 dose of study drug and had SMBG glycemic variability data at the specified time points. Participants were analyzed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles/liter (mmol/L)
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 220 | 221
millimoles/liter (mmol/L)
  SMBG glycemic variability, 12 weeks (n=220, 221) | 2.12 [2.01 to 2.24] | 2.13 [2.01 to 2.24]
  SMBG glycemic variability, 24 weeks (n=216, 216) | 2.03 [1.92 to 2.14] | 1.99 [1.88 to 2.10]

7. Secondary Outcome: Daily Insulin Dose: Total, Basal, and Prandial at 12 Weeks and 24 Weeks
Time Frame: 12 weeks, 24 weeks
Population: Intention-to-treat population (ITT): randomized participants who received at least 1 dose of study drug and had dosing data at the specified time points. Participants were analyzed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Mean (Standard Deviation); unit: international units (IU)
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 236 | 240
international units (IU)
  Total Insulin Dose at 12 Weeks (n=224, 224) | 51.2 (23.60) [32.0 to 65.2] | 49.2 (20.89) [33.0 to 63.3]
  Total Insulin Dose at 24 Weeks LOCF (n=236, 240) | 53.1 (24.60) [34.0 to 68.0] | 50.8 (21.96) [34.0 to 66.0]
  Basal Insulin Dose at 12 Weeks (n=224, 224) | 38.4 (17.70) [24.0 to 48.9] | 37.1 (18.34) [22.0 to 49.5]
  Basal Insulin Dose at 24 Weeks LOCF (n=236, 240) | 39.8 (18.45) [25.5 to 51.0] | 37.4 (18.76) [22.0 to 50.0]
  Prandial Insulin Dose at 12 Weeks (n=224, 224) | 12.8 (5.90) [8.0 to 16.3] | 12.1 (5.10) [8.0 to 16.0]
  Prandial Insulin Dose at 24 Weeks LOCF(n=236, 240) | 13.3 (6.15) [8.5 to 17.0] | 13.5 (6.46) [8.0 to 17.2]

8. Secondary Outcome: Change in Weight From Baseline to 12 Weeks and 24 Weeks
Description: The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included baseline weight as a covariate, treatment, country, baseline glycosylated hemoglobin A1c (HbA1c) stratification level, week of visit, and the treatment-by-week interaction as fixed effects, and participant and error as random effects.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Safety population: randomized participants who took at least 1 dose of study drug and had evaluable body weight data at the specified time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (kg)
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 224 | 225
kilograms (kg)
  Change at 12 weeks (n=224, 225) | 0.54 [0.25 to 0.83] | 0.34 [0.05 to 0.62]
  Change at 24 weeks (n=219, 217) | 1.13 [0.75 to 1.52] | 0.50 [0.11 to 0.89]
Statistical Analysis 1: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.2833, Mixed Models Analysis — p-value is for the comparison at Week 12
Statistical Analysis 2: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; p = 0.0176, Mixed Models Analysis — p-value is for the comparison at Week 24

9. Secondary Outcome: The Number of Participants With a Hypoglycemic Episodes (Incidence)
Description: A hypoglycemic episode was defined as an event associated with 1) reported signs and symptoms of hypoglycemia, and/or 2) a documented blood glucose (BG) concentration of <= 70 milligrams per deciliter [mg/dL, 3.9 millimoles per liter (mmol/L)].
Time Frame: Baseline through 24 weeks
Population: Safety population: randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 236 | 240
participants | 144 | 150

10. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) Score at 24 Weeks
Description: ITSQ: validated instrument containing 22 items which are measured on a 7-point scale: 1 (no bother at all) to 7 (a tremendous bother) used to assess insulin treatment satisfaction. Items are divided into 5 domains: Inconvenience of Regimen (5 items: domain score range 5 to 35), Lifestyle Flexibility (3 items: domain score range 3 to 21), Glycemic Control (3 items: domain score range 3 to 21), Hypoglycemic Control (5 items: domain score range 5 to 35), Insulin Delivery Device (6 items: domain score range 6 to 42) lower scores reflect better outcome. ITSQ Total Overall Score ranged from 22 to 154. Raw domain scores transformed on 0-100 scale, where transformed domain score = 100×[(7-raw domain score)/6]. Higher scores indicate better treatment satisfaction. Least squares (LS) mean estimated from analysis of covariance (ANCOVA) model that included baseline score as covariate and treatment, glycosylated hemoglobin A1c (HbA1c) stratum, and country as fixed effects.
Time Frame: 24 weeks
Population: Randomized participants who received at least 1 dose of study drug and had ITSQ scores at 24 weeks. Last observation carried forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 230 | 229
units on a scale | 80.91 [79.02 to 82.81] | 81.84 [79.97 to 83.72]

11. Secondary Outcome: Perceptions About Medications-Diabetes 21 (PAM-D21) Questionnaire Score at 24 Weeks
Description: PAM-D21 is a validated questionnaire consisting of 21 items to assess a participant's perceptions about their diabetes treatment regimens and perceived emotional and physical side-effects. The PAM-D21 consists of 4 subscales: Convenience/Flexibility (items 1 to 3); Perceived Effectiveness (items 4 to 6); Emotional Effects (items 7 to 11); and Physical Effects (items 12 to 21). Item scores range from 1 (none of the time) to 4 (all of the time). Subscale scores were linearly transformed to a 0-100, with higher score corresponds to better perceptions about diabetes medications. The least squares (LS) mean was estimated from an analysis of covariance (ANCOVA) model that included baseline score as a covariate and treatment, glycosylated hemoglobin A1c (HbA1c) stratum, and country as fixed effects.
Time Frame: 24 weeks
Population: Randomized participants who received at least 1 dose of study drug and had PAM-D21 scores at 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 231 | 230
units on a scale
  Convenience/Flexibility (n= 231, 230) | 83.90 [81.00 to 86.80] | 84.13 [81.26 to 87.00]
  Perceived Effectiveness (n=231, 230) | 76.78 [73.32 to 80.23] | 78.76 [75.34 to 82.17]
  Emotional Effects (n=231, 230) | 81.84 [78.87 to 84.80] | 81.86 [78.92 to 84.79]
  Physical Effects (n=231, 228) | 87.89 [86.20 to 89.58] | 89.04 [87.37 to 90.72]

12. Secondary Outcome: The Rate of Hypoglycemic Episodes
Description: The hypoglycemia rate per 30 days was calculated as the number of episodes reported for the interval between visits and during the study divided by the number of days in the given interval and multiplied by 30.
Time Frame: Baseline through 24 weeks
Population: Safety population: randomized participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: hypoglycemic episodes per 30 day period
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 236 | 240
hypoglycemic episodes per 30 day period | 1.07 (1.181) | 1.36 (2.172)

13. Secondary Outcome: The Number of Participants With Severe Hypoglycemic Episodes
Description: The number of participants who had a severe hypoglycemic episode anytime during the study. Severe hypoglycemia was defined as any event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline through 24 weeks
Population: Safety population: randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 236 | 240
participants | 2 | 0

14. Primary Outcome: Change in HbA1c From Baseline to 24 Weeks Endpoint (Intention-to-Treat Population)
Description: as for outcome 1
Time Frame: Baseline, 24 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Number analyzed (Participants) | 220 | 220
percentage of HbA1c | -1.30 [-1.44 to -1.16] | -1.08 [-1.22 to -0.94]
Statistical Analysis 1: Comparison: Insulin Lispro Low Mixture vs Insulin Glargine+Insulin Lispro; Test type: Superiority or Other; Superiority will be concluded if of 95% CI upper limit for treatment difference (2x-daily insulin lispro LM minus the comparator arm) at 24 wks is <0%; LS mean difference = -0.22, 95% CI 2-sided [-0.39 to -0.05]

ADVERSE EVENTS:
Arm/Group | Insulin Lispro Low Mixture | Insulin Glargine+Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 11/236 | 8/240
Other Adverse Events (participants affected / at risk) | 109/236 | 93/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro Low Mixture (N=236) | Insulin Glargine+Insulin Lispro (N=240)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro Low Mixture (N=236) | Insulin Glargine+Insulin Lispro (N=240)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4)
Apical granuloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Discomfort (General disorders) | 1 (1) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (4)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 4 (4)
Keratitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 20 (24) | 13 (13)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (2)
Respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 3 (4) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4) | 5 (7)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6) | 4 (6)
Headache (Nervous system disorders) | 7 (9) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0/120 (0) | 1/142 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pityriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (4)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Vein disorder (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days